CLINICAL TRIAL: NCT00294827
Title: Liver Transplantation and Metastatic Colo-rectal Cancer.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Smedman, MD, Consultant, gastrointestinal oncology, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-05409 (SECA I)
Record Dates: First submitted 2006-02-21; First posted 2006-02-22 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Colo-rectal Cancer
Keywords: Liver transplantation
MeSH Terms: conditions — Colonic Neoplasms | interventions — Liver Transplantation

ARMS (1):
- Liver transplantation (Experimental)
  Interventions: Procedure: Liver transplantation and colo-rectal cancer

INTERVENTIONS:
Procedure: Liver transplantation and colo-rectal cancer — Liver transplantation

SUMMARY:
Survival of colo-rectal cancer patients after liver transplantation.

DETAILED DESCRIPTION:
Survival, time to progression, other malignancy, side-effects, quality of life.

ELIGIBILITY:
Inclusion Criteria:Colo-rectal cancer -

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2006-02; Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Survival | 6 years

SECONDARY OUTCOMES:
Time to progression side-effects | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Svein Dueland, MD, PhD, Principal Investigator — Rikshospitalet-Radiumhospitalet RRHF
Locations (1):
- Rikshospitalet-Radiumhospitalet HF, Oslo, Norway

REFERENCES:
- [Derived] Foss A, Adam R, Dueland S. Liver transplantation for colorectal liver metastases: revisiting the concept. Transpl Int. 2010 Jul;23(7):679-85. doi: 10.1111/j.1432-2277.2010.01097.x. Epub 2010 Apr 30. PMID 20477993